CLINICAL TRIAL: NCT01646021
Title: A Randomized, Controlled, Open-Label, Multicenter Phase 3 Study of the Bruton's Tyrosine Kinase (BTK) Inhibitor, Ibrutinib, Versus Temsirolimus in Subjects With Relapsed or Refractory Mantle Cell Lymphoma Who Have Received at Least One Prior Therapy
Brief Title: Study of Ibrutinib (a Bruton's Tyrosine Kinase Inhibitor), Versus Temsirolimus in Patients With Relapsed or Refractory Mantle Cell Lymphoma Who Have Received at Least One Prior Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Collaborators: Pharmacyclics LLC. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR100848; PCI-32765MCL3001 (Other: Janssen Research & Development, LLC); 2012-000601-74 (EudraCT Number); U1111-1135-6930 (Other: Universal Trial Number)
Record Dates: First submitted 2012-07-18; First posted 2012-07-20 (Estimated); Results first posted 2017-03-01 (Actual); Last update posted 2018-01-19 (Actual); Status verified 2017-12

CONDITIONS: Mantle Cell Lymphoma
Keywords: Mantle cell lymphoma; Relapsed mantle cell lymphoma; Refractory mantle cell lymphoma; Ibrutinib; Bruton's tyrosine kinase inhibitor; Temsirolimus
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — ibrutinib; temsirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (2):
- Ibrutinib (Experimental)
  Interventions: Drug: Ibrutinib
- Temsirolimus (Experimental)
  Interventions: Drug: Temsirolimus

INTERVENTIONS:
Drug: Ibrutinib — 560 mg once daily continuous (without interruption) by mouth for 21-day cycles
  Arms: Ibrutinib
Drug: Temsirolimus — 175 mg once daily intravenous infusion on Days 1, 8, 15 of the first cycle followed by 75 mg on Days 1, 8, 15 of each 21-day cycle
  Arms: Temsirolimus

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of ibrutinib versus temsirolimus in patients with relapsed or refractory mantle cell lymphoma who received at least 1 prior chemotherapy regimen.

DETAILED DESCRIPTION:
This is a randomized (individuals assigned to study treatment by chance), open-label (identity of assigned study drug will be known), study to evaluate the efficacy and safety of ibrutinib when compared with temsirolimus in patients with relapsed or refractory mantle cell lymphoma (MCL) who have received at least 1 prior rituximab-containing chemotherapy regimen. Approximately 280 eligible patients will be randomly assigned in a 1:1 ratio and stratified (grouped) by the number of prior lines of therapy (1 or 2 versus >=3) and simplified MCL International Prognostic Index criteria to receive either ibrutinib by mouth (Treatment Arm A) or temsirolimus intravenous infusion (Treatment Arm B). The study will consist of screening, treatment, and posttreatment phases. Data will be collected on disease response to the treatment, progression-free survival, overall survival, subsequent anti-MCL therapies, patient reported outcomes, and medical resource utilization. Tumor samples, blood collected at multiple time points, and a bone marrow aspirate will be evaluated to identify markers predictive of response or resistance to ibrutinib. Serial pharmacokinetic (study of what the body does to a drug) samples will be collected as detailed in the protocol. Safety will be monitored throughout the study. Disease evaluations will be performed every 9 weeks for up to 15 months from the start of study drug, and every 24 weeks thereafter, until disease progression, death, or the clinical cutoff, whichever comes first. Patients who receive treatment with temsirolimus and have disease progression (confirmed by an Independent Review Committee) may be eligible to crossover and receive treatment with ibrutinib 560 mg orally, daily, on a 21-day cycle until disease progression, unacceptable toxicity, or study end. Data will be analyzed up to 3 years after the last patient is enrolled for the final follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of mantle cell lymphoma (MCL)
* Received at least 1 prior rituximab-containing chemotherapy regimen (separate lines of therapy are defined as single or combination therapies that are either separated by disease progression or by a > 6 month treatment-free interval)
* Documented relapse or disease progression following the last anti-MCL treatment
* At least 1 measurable site of disease according to Revised Response Criteria for Malignant Lymphoma
* Eastern Cooperative Oncology Group performance status grade 0 or 1
* Protocol-defined hematology and biochemistry laboratory values

Exclusion Criteria:

* Prior nitrosoureas within 6 weeks, chemotherapy within 3 weeks, therapeutic anticancer antibodies within 4 weeks, radio- or toxin-immunoconjugates within 10 weeks, radiation therapy or other investigational agents within 3 weeks, or major surgery within 4 weeks of randomization
* Prior treatment with temsirolimus, other mTOR inhibitors, ibrutinib, or other Bruton's tyrosine kinase (BTK) inhibitors
* Known central nervous system lymphoma
* Received an allogeneic or autologous hematopoietic stem cell transplant <=6 months from the date of randomization and on immunosuppressive therapy or have evidence of active graft versus host disease
* Diagnosed or treated for malignancy other than MCL, except: malignancy treated with curative intent and with no known active disease present for >=3 years before randomization, adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease, adequately treated cervical carcinoma in situ without evidence of disease
* History of stroke or intracranial hemorrhage within 6 months prior to randomization
* Requires anticoagulation with warfarin or equivalent vitamin K antagonist
* Requires treatment with strong CYP3A inhibitor
* Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of Screening, or any Class 3 (moderate) or Class 4 (severe) cardiac disease as defined by the New York Heart Association Functional Classification
* Known history of human immunodeficiency virus (HIV) or active hepatitis C virus (HCV) or active hepatitis B virus (HBV) infection or any uncontrolled active systemic infection requiring intravenous antibiotics
* Woman who is pregnant or breast-feeding
* Any life-threatening illness, medical condition, or organ system dysfunction which, in the investigator's opinion, could compromise the patient's safety, interfere with the absorption or metabolism of ibrutinib capsules, or put the study outcomes at undue risk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2012-12-10 (Actual); Primary Completion 2015-06-05 (Actual); Study Completion 2016-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (92):
- Belgium (7):
  - Antwerp
  - Bruges
  - Brussels
  - Edegem
  - Ghent
  - Leuven
  - Wilrijk
- Brazil (5):
  - Goiânia
  - Porto Alegre
  - Ribeirão Preto
  - Rio de Janeiro
  - São Paulo
- Canada (3):
  - Edmonton, Alberta
  - Ottawa, Ontario
  - Montreal, Quebec
- Temuco, Chile
- Colombia (2):
  - Bogotá
  - Medellín
- Czechia (2):
  - Brno
  - Prague
- France (4):
  - Mulhouse
  - Paris
  - Pessac
  - Villejuif
- Germany (9):
  - Berlin
  - Cologne
  - Essen
  - Heidelberg
  - Homburg
  - Kiel
  - Mainz
  - München
  - Ulm
- Hungary (4):
  - Budapest
  - Debrecen
  - Pécs
  - Szeged
- Dublin, Ireland
- Mexico (3):
  - Monterrey
  - Oaxaca City
  - Querétaro
- Netherlands (2):
  - Amsterdam
  - Rotterdam
- Poland (7):
  - Brzozów
  - Chorzów
  - Gdansk
  - Krakow
  - Opole
  - Słupsk
  - Wroclaw
- Portugal (3):
  - Coimbra
  - Lisbon
  - Porto
- Russia (10):
  - Chelyabinsk
  - Krasnodar
  - Moscow
  - Nizhny Novgorod
  - Obninsk
  - Rostov-on-Don
  - Saint Petersburg
  - Sochi
  - Syktyvkar
  - Yekaterinburg
- South Korea (2):
  - Goyang-si
  - Seoul
- Spain (5):
  - Barcelona
  - Madrid
  - Palma de Mallorca
  - Salamanca
  - Valencia
- Sweden (5):
  - Gothenburg
  - Lund
  - Stockholm
  - Umeå
  - Uppsala
- Taiwan (3):
  - Tainan
  - Taipei
  - Taoyuan District
- Ukraine (6):
  - Cherkassy
  - Dnipro
  - Donetsk
  - Khmelnitskiy
  - Kiev
  - Lviv
- United Kingdom (8):
  - Birmingham
  - Harrow
  - Leeds
  - Liverpool
  - London
  - Manchester
  - Plymouth
  - Southampton

REFERENCES:
- [Derived] Brown JR, Moslehi J, O'Brien S, Ghia P, Hillmen P, Cymbalista F, Shanafelt TD, Fraser G, Rule S, Kipps TJ, Coutre S, Dilhuydy MS, Cramer P, Tedeschi A, Jaeger U, Dreyling M, Byrd JC, Howes A, Todd M, Vermeulen J, James DF, Clow F, Styles L, Valentino R, Wildgust M, Mahler M, Burger JA. Characterization of atrial fibrillation adverse events reported in ibrutinib randomized controlled registration trials. Haematologica. 2017 Oct;102(10):1796-1805. doi: 10.3324/haematol.2017.171041. Epub 2017 Jul 27. PMID 28751558
- [Derived] Dreyling M, Jurczak W, Jerkeman M, Silva RS, Rusconi C, Trneny M, Offner F, Caballero D, Joao C, Witzens-Harig M, Hess G, Bence-Bruckler I, Cho SG, Bothos J, Goldberg JD, Enny C, Traina S, Balasubramanian S, Bandyopadhyay N, Sun S, Vermeulen J, Rizo A, Rule S. Ibrutinib versus temsirolimus in patients with relapsed or refractory mantle-cell lymphoma: an international, randomised, open-label, phase 3 study. Lancet. 2016 Feb 20;387(10020):770-8. doi: 10.1016/S0140-6736(15)00667-4. Epub 2015 Dec 7. PMID 26673811

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 139 participants were randomized and treated in the ibrutinib arm and 141 participants were randomized to the temsirolimus arm.
Groups:
- Ibrutinib: Participants received 560 milligram (mg) ibrutinib (4*140 mg capsules) by mouth once daily continuous (without interruption) self-administered home treatment during the 21 day cycle.
- Temsirolimus: Participants received Temsirolimus intravenous (IV) infusion 175 mg on Days 1, 8, 15 of the first cycle followed by 75 mg on Days 1, 8, 15 of each subsequent 21 day cycle. Each temsirolimus dose is infused over a 30 to 60 minute period.
Period: Overall Study
Arm/Group | Ibrutinib | Temsirolimus
Started | 139 | 141
Treated | 139 | 139
Completed | 0 | 0
Not Completed | 139 | 141
Not completed — Death | 77 | 83
Not completed — Study Terminated by Sponsor | 50 | 41
Not completed — Lost to Follow-up | 2 | 2
Not completed — Withdrawal by Subject | 10 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ibrutinib | Temsirolimus | Total
Number analyzed (Participants) | 139 | 141 | 280
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 53 | 54 | 107
  >=65 years | 86 | 87 | 173
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.7 (8.68) | 67.1 (9.83) | 66.9 (9.26)
Sex/Gender, Customized [Number; unit: participants]
  Female | 39 | 33 | 72
  Male | 100 | 108 | 208
Region of Enrollment [Number; unit: participants]
  Belgium | 7 | 10 | 17
  Brazil | 5 | 10 | 15
  Canada | 6 | 3 | 9
  Colombia | 3 | 4 | 7
  Czech Republic | 7 | 7 | 14
  Germany | 12 | 11 | 23
  Spain | 5 | 14 | 19
  France | 5 | 5 | 10
  United Kingdom | 11 | 16 | 27
  Hungary | 5 | 7 | 12
  Ireland | 2 | 1 | 3
  Italy | 6 | 8 | 14
  South Korea | 11 | 3 | 14
  Mexico | 1 | 1 | 2
  Netherlands | 2 | 0 | 2
  Poland | 9 | 14 | 23
  Portugal | 3 | 3 | 6
  Russian Federation | 18 | 11 | 29
  Sweden | 10 | 8 | 18
  Taiwan | 5 | 1 | 6
  Ukraine | 6 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the duration in months from the date of randomization to the date of progression disease (PD) or relapse from complete response (CR) or death whichever was reported first and was assessed based on the investigator assessment. Revised Response Criteria for Malignant Lymphoma categorizes the response of the treatment of a patient's tumour to CR (the disappearance of all evidence of disease), Relapsed Disease or PD (Any new lesion or increase by greater than or equal to [>=] 50 percent [%] of previously involved sites from nadir).
Time Frame: Time from the date of randomization until the date of first documented evidence of progressive disease (or relapse for subjects who experience CR during the study) or death, whichever occurred first (approximately 48 months)
Population: The Intent-to-Treat (ITT) population included all participants randomized into the study regardless of treatment actually received.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ibrutinib | Temsirolimus
Number analyzed (Participants) | 139 | 141
Months | 15.6 [10.6 to 25.1] | 6.2 [4.2 to 7.8]
Statistical Analysis 1: Comparison: Ibrutinib vs Temsirolimus; Test type: Other; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.45, 95% CI 2-sided [0.35 to 0.60]

2. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR is defined as the percentage of participants who achieved either CR or PR as best overall response based on the investigator assessment. CR is Disappearance of all target lesions while PR is greater than or equal to 30 % decrease in the sum of the longest diameter of target lesions and Overall Response (OR) is sum of CR and PR.
Time Frame: Approximately up to 48 months
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Ibrutinib | Temsirolimus
Number analyzed (Participants) | 139 | 141
Percentage of participants | 77.0 | 46.8

3. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) was defined as the interval between the date of randomization and the date of death from any cause.
Time Frame: Approximately up to 48 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ibrutinib | Temsirolimus
Number analyzed (Participants) | 139 | 141
Months | 30.3 [19.1 to 42.1] | 23.5 [13.0 to 30.7]
Statistical Analysis 1: Comparison: Ibrutinib vs Temsirolimus; Test type: Superiority; p = 0.0621, Log Rank; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.54 to 1.02]

4. Secondary Outcome: Duration of Response
Description: Duration of response (CR or PR), defined as the duration in days from the date of initial response to the date of first documented evidence of progressive disease (or relapse for participants who experience CR during the study) or death. The analysis was based on the investigator assessment.
Time Frame: Approximately up to 48 months
Population: The Intent-to-Treat (ITT) population included all participants randomized into the study regardless of treatment actually received. The 'N' (number of participants analyzed) signifies the number of participants responded for this outcome measure.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ibrutinib | Temsirolimus
Number analyzed (Participants) | 107 | 66
Months | 23.1 [16.2 to 28.1] | 6.3 [4.7 to 8.6]

5. Secondary Outcome: Time-to-Next Treatment
Description: Time to next treatment was measured from the date of randomization to the start date of any anti-neoplastic treatment subsequent to study treatment.
Time Frame: Approximately up to 48 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ibrutinib | Temsirolimus
Number analyzed (Participants) | 139 | 141
Months | 31.8 [23.3 to NA] — upper 95%CI was not estimable due to less than 50% participants had events occurred | 11.6 [8.0 to 13.3]

6. Secondary Outcome: Progression-Free Survival 2
Description: Progression-free survival 2 defined as the time interval between the date of randomization and date of event, defined as progressive disease as assessed by investigator that started after the next line of subsequent anti-neoplastic therapy (including cross-over to ibrutinib), death from any cause, or the start of the second subsequent anti-neoplastic therapy if no progressive disease was recorded after the first subsequent anti-neoplastic therapy.
Time Frame: Approximately up to 48 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ibrutinib | Temsirolimus
Number analyzed (Participants) | 139 | 141
Months | 26.2 [17.2 to 32.4] | 15.4 [10.2 to 21.3]

7. Secondary Outcome: Time to Worsening in the Lymphoma Sub Scale of Functional Assessment of Cancer Therapy- Lymphoma (FACT-Lym)
Description: Time to worsening in the Lymphoma subscale of the FACT-Lym, defined as the interval from the date of randomization to the start date of worsening. Worsening was defined by a 5-point decrease from baseline. FACT-Lym Lymphoma subscale contains 15 questions, scores from 0 to 4 for each question (higher the worse). Lymphoma subscale score is the total of reverse scores, range 0 to 60. Higher scores indicate a better quality of life.
Time Frame: Approximately up to 48 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Ibrutinib | Temsirolimus
Number analyzed (Participants) | 139 | 141
Weeks | NA [81.4 to NA] — Here, NA indicates median and upper limit of CI of FACT-Lym was not estimable at final analysis due to less than 50% patients had events occurred. | 10.6 [6.6 to 15.3]

8. Secondary Outcome: Number of Participants Affected With Treatment-emergent Adverse Events
Description: An AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Time from first dose of study drug until the last dose date + 30 days or the start of a subsequent anti-neoplastic therapy, whichever occur earlier (Approximately up to 4 years)
Population: Safety population included all randomized participants who received at least 1 dose of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrutinib | Temsirolimus
Number analyzed (Participants) | 139 | 139
Participants | 139 | 138

9. Other Pre Specified Outcome: Time to Response
Description: Time to response for participants with CR/PR, defined as the interval between the date of randomization and date of initial documentation of response.
Time Frame: Approximately up to 2.8 years
Population: as for outcome 4
Measure: Median (Full Range); unit: Months
Arm/Group | Ibrutinib | Temsirolimus
Number analyzed (Participants) | 100 | 57
Months | 2.15 [0.5 to 10.4] | 2.14 [0.9 to 12.0]

10. Other Pre Specified Outcome: Extent of Exposure of Time
Description: Extent of exposure is defined as the duration of the treatment administered during the study. Duration of exposure is calculated as the number of months between the start and end of treatment.
Time Frame: Approximately up to 46.8 months
Population: Safety Analyses Set (SAS) population includes all the randomized participants who received at least 1 dose of study agent (ibrutinib or temsirolimus) during the treatment phase.
Measure: Median (Full Range); unit: Months
Arm/Group | Ibrutinib | Temsirolimus
Number analyzed (Participants) | 139 | 139
Months | 14.39 [0.0 to 46.8] | 3.02 [0.0 to 31.4]

11. Other Pre Specified Outcome: One Year Survival Rate
Description: One -year survival rate, defined as the proportion of participants who were alive 1 year after randomization.
Time Frame: Month 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Ibrutinib | Temsirolimus
Number analyzed (Participants) | 139 | 141
Proportion of participants | 0.68 [0.59 to 0.75] | 0.61 [0.52 to 0.69]

12. Other Pre Specified Outcome: Area Under the Plasma Concentration of Ibrutinib During Steady State (AUC-ss)
Description: The AUC-ss is the area under the plasma concentration time curve observed during steady state.
Time Frame: Cycle 1 and 2 (Day 1): Predose, 1, 2, 4 hr. postdose; Cycle 3 (day 1): Predose (Each cycle is of 21 days)
Population: Pharmacokinetic analysis set included the participants who had received one dose of study drug had at least 1 pharmacokinetic sample obtained post-treatment.
Measure: Mean (Standard Deviation); unit: nanogram*hour per milliliter (ng*h/mL)
Arm/Group | Ibrutinib
Number analyzed (Participants) | 139
nanogram*hour per milliliter (ng*h/mL) | 561.6 (448)

13. Other Pre Specified Outcome: Number of Participants With Biomarkers That Alter B-cell Receptor (BCR) Signaling or Activate Alternative Signaling Pathways and to Explore Their Association With Response or Resistance to Ibrutinib
Description: Biomarker evaluations to identify markers altering BCR signaling or activate alternative signaling pathways and explore their association with response or resistance to ibrutinib. Next-generation sequencing at baseline identifies possible primary resistance mutations and those found only at progression are acquired mutations on therapy.
Time Frame: Approximately up to 28.2 months
Measure: Number; unit: Participants
Arm/Group | Ibrutinib | Temsirolimus
Number analyzed (Participants) | 139 | 141
Participants | 61 | 53

14. Other Pre Specified Outcome: Number of Hospitalizations Reported Related Medical Resource Utilization Information (MRUI)
Description: Medical resource utilization data associated with medical encounters related to disease was reported for all participants throughout the study.
Time Frame: Approximately up to 28.2 months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Hospitalizations
Arm/Group | Ibrutinib | Temsirolimus
Number analyzed (Participants) | 83 | 91
Hospitalizations | 3.1 (4.6) | 2.8 (4.3)

15. Other Pre Specified Outcome: Number of Emergency Room Visits Reported Related Medical Resource Utilization Information (MRUI)
Description: as for outcome 14
Time Frame: Approximately up to 28.2 months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Emergency room visits
Arm/Group | Ibrutinib | Temsirolimus
Number analyzed (Participants) | 5 | 5
Emergency room visits | 1.2 (0.4) | 1.2 (0.4)

16. Other Pre Specified Outcome: Days of Hospitalization and Emergency Room Visits Reported Related Medical Resource Utilization Information (MRUI)
Description: as for outcome 14
Time Frame: Approximately up to 28.2 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Ibrutinib | Temsirolimus
Number analyzed (Participants) | 139 | 141
Days
  Mean days of hospitalization: number analyzed (Participants) | 83 | 91
  Mean days of hospitalization | 19.7 (20.5) | 20.3 (22.4)
  Mean days of emergency room visits: number analyzed (Participants) | 5 | 5
  Mean days of emergency room visits | 1.8 (1.3) | 1.6 (1.3)

17. Other Pre Specified Outcome: The Mean Change From Baseline in Euro QoL Five-Dimension (EQ-5D-5L) Scores for Each Post Baseline Assessment
Description: The EQ-5D is a participant rated questionnaire to assess health-related quality of life in terms of a single utility score. Health State Profile component assesses level of current health for 5 domains: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression, using 5 levels (1=no problems, 2=slight problems, 3=moderate problems, 4=severe problems, and 5=extreme problems). Scoring formula developed by EuroQol Group assigns a utility value for each domain in the profile. Score is transformed and possible total score range -0.594 to 1; higher score indicates a better health state.
Time Frame: Baseline, Cycle 2, 3, 4, 5, 6, 7, 8, 11, 14, 17, 20, 28, 36 and End of treatment (approximately up to 23 months)
Population: The Intent-to-Treat (ITT) population included all participants randomized into the study regardless of treatment actually received. The 'N' (number of participants analyzed) signifies the number of participants evaluated for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Ibrutinib | Temsirolimus
Number analyzed (Participants) | 138 | 130
Units on scale
  Baseline: number analyzed (Participants) | 130 | 120
  Baseline | 0.7 (0.2) | 0.7 (0.2)
  Change at Cycle 2: number analyzed (Participants) | 113 | 95
  Change at Cycle 2 | 0.0 (0.2) | 0.0 (0.2)
  Change at Cycle 3: number analyzed (Participants) | 115 | 85
  Change at Cycle 3 | 0.1 (0.2) | -0.1 (0.2)
  Change at Cycle 4: number analyzed (Participants) | 103 | 70
  Change at Cycle 4 | 0.0 (0.2) | 0.0 (0.3)
  Change at Cycle 5: number analyzed (Participants) | 102 | 57
  Change at Cycle 5 | 0.0 (0.2) | 0.0 (0.2)
  Change at Cycle 6: number analyzed (Participants) | 99 | 49
  Change at Cycle 6 | 0.1 (0.2) | 0.0 (0.2)
  Change at Cycle 7: number analyzed (Participants) | 98 | 39
  Change at Cycle 7 | 0.0 (0.2) | 0.0 (0.2)
  Change at Cycle 8: number analyzed (Participants) | 90 | 37
  Change at Cycle 8 | 0.0 (0.2) | 0.0 (0.2)
  Change at Cycle 11: number analyzed (Participants) | 88 | 33
  Change at Cycle 11 | 0.0 (0.2) | 0.0 (0.2)
  Change at Cycle 14: number analyzed (Participants) | 72 | 26
  Change at Cycle 14 | 0.0 (0.2) | 0.0 (0.1)
  Change at Cycle 17: number analyzed (Participants) | 69 | 19
  Change at Cycle 17 | 0.0 (0.2) | 0.0 (0.2)
  Change at Cycle 20: number analyzed (Participants) | 64 | 16
  Change at Cycle 20 | 0.0 (0.2) | 0.0 (0.2)
  Change at Cycle 28: number analyzed (Participants) | 22 | 6
  Change at Cycle 28 | -0.1 (0.2) | 0.1 (0.2)
  Change at Cycle 36: number analyzed (Participants) | 10 | 4
  Change at Cycle 36 | 0.0 (0.3) | -0.1 (0.2)
  Change at End of treatment: number analyzed (Participants) | 23 | 65
  Change at End of treatment | 0.0 (0.2) | -0.1 (0.3)

ADVERSE EVENTS:
Time Frame: Approximately up to 4 years
Description: Safety population included all randomized participants who received at least 1 dose of study agent (ibrutinib or temsirolimus) during the treatment phase.
Arm/Group | Ibrutinib | Temsirolimus
All-Cause Mortality (participants affected / at risk) | 130/139 | 137/139
Serious Adverse Events (participants affected / at risk) | 79/139 | 83/139
Other Adverse Events (participants affected / at risk) | 130/139 | 137/139
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ibrutinib (N=139) | Temsirolimus (N=139)
Anaemia (Blood and lymphatic system disorders) | 4 | 5
Autoimmune Haemolytic Anaemia (Blood and lymphatic system disorders) | 1 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 2 | 1
Leukocytosis (Blood and lymphatic system disorders) | 2 | 0
Lymphocytosis (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 1
Splenic Infarction (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 3
Acute Myocardial Infarction (Cardiac disorders) | 1 | 0
Angina Pectoris (Cardiac disorders) | 0 | 1
Angina Unstable (Cardiac disorders) | 0 | 1
Arteriosclerosis Coronary Artery (Cardiac disorders) | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 7 | 2
Atrial Flutter (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0
Cardiac Arrest (Cardiac disorders) | 0 | 1
Cardiac Failure Acute (Cardiac disorders) | 0 | 1
Cardiac Failure Chronic (Cardiac disorders) | 1 | 1
Cardiac Failure Congestive (Cardiac disorders) | 0 | 1
Cardiopulmonary Failure (Cardiac disorders) | 0 | 1
Coronary Artery Insufficiency (Cardiac disorders) | 1 | 0
Coronary Artery Stenosis (Cardiac disorders) | 0 | 1
Myocardial Ischaemia (Cardiac disorders) | 0 | 1
Pericarditis (Cardiac disorders) | 1 | 0
Supraventricular Tachycardia (Cardiac disorders) | 1 | 0
Cataract (Eye disorders) | 0 | 1
Diabetic Retinopathy (Eye disorders) | 1 | 0
Vitreous Haemorrhage (Eye disorders) | 1 | 0
Abdominal Hernia (Gastrointestinal disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 5 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 4
Duodenal Stenosis (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Gastric Ulcer (Gastrointestinal disorders) | 1 | 0
Gastritis Haemorrhagic (Gastrointestinal disorders) | 0 | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Intestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Proctitis (Gastrointestinal disorders) | 1 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 3
Vomiting (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 2 | 3
General Physical Health Deterioration (General disorders) | 3 | 5
Malaise (General disorders) | 0 | 1
Mucosal Inflammation (General disorders) | 0 | 1
Multi-Organ Failure (General disorders) | 4 | 0
Oedema (General disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 3 | 7
Hepatitis Toxic (Hepatobiliary disorders) | 1 | 1
Hypersensitivity (Immune system disorders) | 0 | 1
Abscess Limb (Infections and infestations) | 1 | 0
Atypical Pneumonia (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 0
Bronchopulmonary Aspergillosis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Clostridium Difficile Colitis (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 0 | 1
Device Related Infection (Infections and infestations) | 1 | 2
Diverticulitis (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 2
Hepatitis B (Infections and infestations) | 1 | 0
Herpes Zoster (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 1 | 2
Infectious Colitis (Infections and infestations) | 0 | 1
Laryngitis (Infections and infestations) | 1 | 0
Laryngitis Fungal (Infections and infestations) | 0 | 1
Liver Abscess (Infections and infestations) | 0 | 1
Lower Respiratory Tract Infection (Infections and infestations) | 2 | 1
Lung Infection (Infections and infestations) | 2 | 2
Neutropenic Sepsis (Infections and infestations) | 0 | 1
Oral Candidiasis (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 0
Pneumocystis Jirovecii Infection (Infections and infestations) | 0 | 1
Pneumocystis Jirovecii Pneumonia (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 16 | 12
Pneumonia Escherichia (Infections and infestations) | 0 | 1
Pulmonary Tuberculosis (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
Respiratory Tract Infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 6 | 5
Septic Shock (Infections and infestations) | 2 | 1
Sinusitis (Infections and infestations) | 0 | 1
Sinusitis Aspergillus (Infections and infestations) | 0 | 1
Skin Infection (Infections and infestations) | 2 | 1
Soft Tissue Infection (Infections and infestations) | 1 | 0
Tooth Infection (Infections and infestations) | 0 | 1
Tracheitis (Infections and infestations) | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 2
Urinary Tract Infection (Infections and infestations) | 1 | 3
Urinary Tract Infection Bacterial (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Fibula Fracture (Injury, poisoning and procedural complications) | 0 | 1
Foreign Body (Injury, poisoning and procedural complications) | 0 | 1
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 1 | 0
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 2 | 1
Post Procedural Swelling (Injury, poisoning and procedural complications) | 1 | 0
Rib Fracture (Injury, poisoning and procedural complications) | 1 | 0
Splenic Rupture (Injury, poisoning and procedural complications) | 2 | 1
Subdural Haematoma (Injury, poisoning and procedural complications) | 1 | 0
Toxicity to Various Agents (Injury, poisoning and procedural complications) | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 1
Blood Creatinine Increased (Investigations) | 1 | 0
Haemoglobin Decreased (Investigations) | 1 | 0
Neutrophil Count Decreased (Investigations) | 1 | 0
Platelet Count Decreased (Investigations) | 2 | 0
Cachexia (Metabolism and nutrition disorders) | 1 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 2 | 1
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 1
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Tumour Lysis Syndrome (Metabolism and nutrition disorders) | 1 | 3
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Chondrocalcinosis Pyrophosphate (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral Disc Compression (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Adenocarcinoma Gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Laryngeal Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Salivary Gland Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ataxia (Nervous system disorders) | 0 | 1
Cerebral Ischaemia (Nervous system disorders) | 0 | 1
Cerebrovascular Accident (Nervous system disorders) | 0 | 1
Cognitive Disorder (Nervous system disorders) | 1 | 0
Dysarthria (Nervous system disorders) | 2 | 0
Epilepsy (Nervous system disorders) | 1 | 0
Facial Paresis (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Ischaemic Stroke (Nervous system disorders) | 0 | 1
Memory Impairment (Nervous system disorders) | 1 | 0
Myoclonus (Nervous system disorders) | 1 | 0
Neuralgia (Nervous system disorders) | 0 | 2
Syncope (Nervous system disorders) | 1 | 0
Transient Ischaemic Attack (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 0 | 1
Confusional State (Psychiatric disorders) | 1 | 2
Mental Disorder (Psychiatric disorders) | 1 | 0
Acute Kidney Injury (Renal and urinary disorders) | 2 | 1
Cystitis Haemorrhagic (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Nephrotic Syndrome (Renal and urinary disorders) | 1 | 0
Renal Failure (Renal and urinary disorders) | 3 | 4
Renal Impairment (Renal and urinary disorders) | 0 | 1
Pelvic Pain (Reproductive system and breast disorders) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Lung Disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung Infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 6 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Guttate Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0
Panniculitis (Skin and subcutaneous tissue disorders) | 1 | 0
Skin Ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Deep Vein Thrombosis (Vascular disorders) | 0 | 1
Haemorrhage (Vascular disorders) | 2 | 0
Orthostatic Hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ibrutinib (N=139) | Temsirolimus (N=139)
Anaemia (Blood and lymphatic system disorders) | 27 | 57
Neutropenia (Blood and lymphatic system disorders) | 21 | 36
Thrombocytopenia (Blood and lymphatic system disorders) | 25 | 77
Atrial Fibrillation (Cardiac disorders) | 8 | 1
Cataract (Eye disorders) | 2 | 7
Abdominal Pain (Gastrointestinal disorders) | 8 | 11
Abdominal Pain Upper (Gastrointestinal disorders) | 8 | 3
Constipation (Gastrointestinal disorders) | 13 | 21
Diarrhoea (Gastrointestinal disorders) | 45 | 42
Dyspepsia (Gastrointestinal disorders) | 9 | 1
Mouth Ulceration (Gastrointestinal disorders) | 0 | 8
Nausea (Gastrointestinal disorders) | 20 | 30
Oral Pain (Gastrointestinal disorders) | 1 | 9
Stomatitis (Gastrointestinal disorders) | 4 | 28
Vomiting (Gastrointestinal disorders) | 17 | 9
Asthenia (General disorders) | 12 | 26
Fatigue (General disorders) | 31 | 40
Mucosal Inflammation (General disorders) | 2 | 21
Oedema Peripheral (General disorders) | 19 | 33
Pyrexia (General disorders) | 24 | 26
Bronchitis (Infections and infestations) | 8 | 8
Conjunctivitis (Infections and infestations) | 17 | 9
Herpes Zoster (Infections and infestations) | 10 | 5
Nasopharyngitis (Infections and infestations) | 16 | 16
Oral Herpes (Infections and infestations) | 4 | 15
Paronychia (Infections and infestations) | 9 | 5
Pneumonia (Infections and infestations) | 6 | 14
Respiratory Tract Infection (Infections and infestations) | 9 | 14
Rhinitis (Infections and infestations) | 8 | 5
Sinusitis (Infections and infestations) | 11 | 6
Upper Respiratory Tract Infection (Infections and infestations) | 28 | 15
Urinary Tract Infection (Infections and infestations) | 10 | 7
Contusion (Injury, poisoning and procedural complications) | 10 | 3
Alanine Aminotransferase Increased (Investigations) | 4 | 9
Aspartate Aminotransferase Increased (Investigations) | 5 | 10
Blood Alkaline Phosphatase Increased (Investigations) | 4 | 9
Blood Creatinine Increased (Investigations) | 16 | 18
Blood Lactate Dehydrogenase Increased (Investigations) | 2 | 7
Neutrophil Count Decreased (Investigations) | 7 | 10
Platelet Count Decreased (Investigations) | 11 | 23
Weight Decreased (Investigations) | 9 | 18
Decreased Appetite (Metabolism and nutrition disorders) | 26 | 25
Diabetes Mellitus (Metabolism and nutrition disorders) | 1 | 7
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 | 18
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 26
Hyperkalaemia (Metabolism and nutrition disorders) | 9 | 3
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 25
Hypokalaemia (Metabolism and nutrition disorders) | 12 | 24
Hypomagnesaemia (Metabolism and nutrition disorders) | 9 | 4
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 9
Back Pain (Musculoskeletal and connective tissue disorders) | 15 | 14
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 26 | 4
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 5 | 12
Dysgeusia (Nervous system disorders) | 1 | 7
Headache (Nervous system disorders) | 13 | 17
Insomnia (Psychiatric disorders) | 7 | 15
Cough (Respiratory, thoracic and mediastinal disorders) | 31 | 31
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 | 13
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 13 | 31
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 8 | 8
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 10 | 5
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 7
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 12 | 18
Rash (Skin and subcutaneous tissue disorders) | 18 | 25
Rash Generalised (Skin and subcutaneous tissue disorders) | 1 | 7
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 5 | 7
Skin Lesion (Skin and subcutaneous tissue disorders) | 6 | 8
Haematoma (Vascular disorders) | 11 | 3
Hypertension (Vascular disorders) | 16 | 5
Hypotension (Vascular disorders) | 7 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.